CLINICAL TRIAL: NCT04223778
Title: A Phase 3 Randomized, Active-Controlled, Open-Label Clinical Study to Evaluate a Switch to Doravirine/Islatravir (DOR/ISL) Once-Daily in Participants With HIV-1 Virologically Suppressed on Antiretroviral Therapy
Brief Title: Safety and Efficacy of a Switch to Doravirine/Islatravir in Participants With HIV-1 (MK-8591A-017)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8591A-017; MK-8591A-017 (Other: MSD); 205165 (Registry Identifier: JAPIC-CTI); 2019-000586-20 (EudraCT Number)
Record Dates: First submitted 2020-01-08; First posted 2020-01-10 (Actual); Results first posted 2022-09-19 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Doravirine/Islatravir (DOR/ISL) (Experimental): Participants who were previously treated with continuous baseline antiretroviral therapy (ART) will receive DOR/ISL, a fixed dose combination (FDC) of 100 mg doravirine (DOR)/0.75 mg islatravir (ISL) orally once daily for 96 weeks.
  Interventions: Drug: DOR/ISL
- Group 2: Baseline Antiretroviral Therapy (ART) (Active Comparator): Participants received continuous baseline ART for 48 weeks. Continuing participants delayed switch over from baseline ART to DOR/ISL, fixed dose combination of 100 mg DOR/0.75 mg ISL orally once daily, from Week 48 to Week 96, a total DOR/ISL treatment duration of 48 Weeks.
  Interventions: Drug: DOR/ISL; Drug: ART

INTERVENTIONS:
Drug: DOR/ISL — A FDC of 100 mg DOR/ 0.75 mg ISL taken in tablet form, orally, once daily
  Other Names: MK-8591A
Drug: ART — Baseline ART regimen will be administered as per approved label. ART medication will not be provided by the Sponsor; participants will provide their own ART medications. Allowed drug classes include nucleoside analog reverse transcriptase inhibitors (NRTIs), non-nucleoside reverse transcriptase inhibitors (NNRTIs), protease inhibitors (PIs), integrase strand transferase inhibitors (InSTIs), fusion inhibitors, chemokine receptor 5 (CCR5) antagonists, post-attachment inhibitor, and pharmacokinetic (PK) boosters.
  Arms: Group 2: Baseline Antiretroviral Therapy (ART)

SUMMARY:
This study will evaluate the safety and efficacy of a switch to MK-8591A (a fixed dose combination of doravirine and islatravir) in human immunodeficiency virus -1 (HIV-1)-infected participants virologically suppressed on a protocol-specified antiretroviral regimen. The primary hypothesis is that a switch to MK-8591A will be non-inferior to continued treatment with baseline antiretroviral therapy (ART) as assessed by the percentage of participants with HIV-1 ribonucleic acid (RNA) ≥50 copies/mL at Week 48.

ELIGIBILITY:
Inclusion Criteria:

* Is human immunodeficiency virus (HIV-1) positive
* Has been receiving continuous, stable oral 2-drug or 3-drug combination (± pharmacokinetic (PK) booster) with documented viral suppression (HIV-1 RNA <50 copies/mL) for ≥3 months prior to signing informed consent and has no history of prior virologic treatment failure on any past or current regimen.
* Females are eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: is not a woman of childbearing potential (WOCBP); is a WOCBP and using an acceptable contraceptive method, or be abstinent from heterosexual intercourse as their preferred and usual lifestyle; a WOCBP must have a negative highly sensitive pregnancy test ([urine or serum] as required by local regulations) within 24 hours before the first dose of study intervention; if a urine test cannot be confirmed as negative (e.g. an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive

Exclusion Criteria:

* Has HIV-2 infection
* Has hypersensitivity or other contraindication to any of the components of the study interventions as determined by the investigator
* Has an active diagnosis of hepatitis due to any cause, including active Hepatitis B Virus (HBV) co-infection
* Has a history of malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or cutaneous Kaposi's sarcoma
* Is taking or is anticipated to require systemic immunosuppressive therapy, immune modulators, or any prohibited therapies
* Is currently taking long-acting cabotegravir-rilpivirine
* Is currently participating in or has participated in a clinical study with an investigational compound or device from 45 days prior to Day 1 through the study treatment period
* Has a documented or known virologic resistance to doravirine (DOR)
* Expects to conceive or donate eggs at any time during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 672 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2024-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (78):
- United States (15):
  - Georgetown University Hospital ( Site 1018), Washington D.C., District of Columbia
  - Midway Immunology and Research ( Site 1030), Ft. Pierce, Florida
  - Orlando Immunology Center ( Site 1007), Orlando, Florida
  - Bliss Healthcare Services ( Site 1025), Orlando, Florida
  - Triple O Research Institute, P.A. ( Site 1026), West Palm Beach, Florida
  - Chatham County Health Department ( Site 1043), Savannah, Georgia
  - Northstar Healthcare ( Site 1002), Chicago, Illinois
  - Kansas City CARE Health Center ( Site 1008), Kansas City, Missouri
  - ID Care ( Site 1023), Hillsborough, New Jersey
  - University of North Carolina at Chapel Hill ( Site 1042), Chapel Hill, North Carolina
  - University of Pennsylvania ( Site 1038), Philadelphia, Pennsylvania
  - Saint Hope Foundation, Inc. ( Site 1037), Bellaire, Texas
  - North Texas ID Consultants, PA ( Site 1003), Dallas, Texas
  - Texas Centers for Infectious Disease Associates P.A. ( Site 1022), Fort Worth, Texas
  - The Crofoot Research Center, Inc. ( Site 1005), Houston, Texas
- Australia (4):
  - Holdsworth House Medical Practice ( Site 2300), Sydney, New South Wales
  - Royal Brisbane and Womens Hospital- Infectious Diseases Unit ( Site 2309), Herston, Queensland
  - Melbourne Sexual Health Centre ( Site 2305), Carlton, Victoria
  - Fiona Stanley Hospital ( Site 2301), Murdoch, Western Australia
- Canada (7):
  - Southern Alberta HIV Clinic ( Site 1108), Calgary, Alberta
  - Vancouver ID Research and Care Centre Society ( Site 1100), Vancouver, British Columbia
  - Hamilton Health Sciences ( Site 1103), Hamilton, Ontario
  - Maple Leaf Research ( Site 1112), Toronto, Ontario
  - Toronto General Hospital - University Health Network ( Site 1105), Toronto, Ontario
  - Clinique de Medecine Urbaine du Quartier Latin ( Site 1104), Montreal, Quebec
  - Clinique Medicale L Actuel ( Site 1114), Montreal, Quebec
- Chile (3):
  - Hospital Dr. Hernan Henriquez Aravena ( Site 1305), Temuco, Región de la Araucanía
  - Clinica Arauco Salud ( Site 1300), Santiago, Santiago Metropolitan
  - Centro de Investigacion Clinica UC CICUC ( Site 1303), Santiago, Santiago Metropolitan
- Fundacion Valle del Lili ( Site 1201), Cali, Valle del Cauca Department, Colombia
- France (7):
  - Hopital de la Croix-Rousse ( Site 2027), Lyon, Auvergne-Rhône-Alpes
  - Hopital Francois Mitterrand ( Site 2019), Dijon, Cote-d'Or
  - CHU de Bordeaux- Hopital Saint Andre ( Site 2015), Bordeaux, Gironde
  - CHU de Toulouse - Hopital Purpan ( Site 2004), Toulouse, Haute-Garonne
  - CHU Hotel Dieu Nantes ( Site 2020), Nantes, Loire-Atlantique
  - CHU de Rouen ( Site 2005), Rouen, Seine-Maritime
  - A.P.H. Paris, Hopital Saint Louis ( Site 2014), Paris
- Italy (3):
  - ASST Fatebenefratelli-Ospedale Sacco ( Site 2200), Milan
  - A.O.U. Universita degli Studi della Campania-Luigi Vanvitelli ( Site 2208), Napoli
  - Policlinico Gemelli Instituto di Clinica Chirurgica ( Site 2206), Roma
- Japan (5):
  - National Hospital Organization Nagoya Medical Center ( Site 2403), Nagoya, Aichi-ken
  - National Hospital Organization Osaka National Hospital ( Site 2402), Osaka
  - Tokyo Metropolitan Komagome Hospital ( Site 2406), Tokyo
  - Tokyo Medical University Hospital ( Site 2404), Tokyo
  - Center Hospital of the National Center for Global Health and Medicine ( Site 2401), Tokyo
- Christchurch Hospital ( Site 2303), Christchurch, Canterbury, New Zealand
- Poland (4):
  - EMC Instytut Medyczny SA Przychodnia przy ul. Lowieckiej we Wroclawiu ( Site 1500), Wroclaw, Lower Silesian Voivodeship
  - SP ZOZ Wojewodzki Szpital Zakazny ( Site 1505), Warsaw, Masovian Voivodeship
  - Wroclawskie Centrum Zdrowia SP ZOZ ( Site 1507), Wroclaw
  - Wojewodzki Szpital Specjalistyczny im. dr. Wladyslawa Bieganskiego ( Site 1503), Lodz-Baluty, Łódź Voivodeship
- Russia (8):
  - Kemerovo Regional Center for the Prevention and Control of AIDS ( Site 1713), Kemerovo, Kemerovo Oblast
  - Krasnoyarsk Regional Center for Prevention and Control of AIDS ( Site 1712), Krasnoyarsk, Krasnoyarsk Krai
  - Saint Petersburg Center for Prophylactic of AIDS and Inf. Diseases ( Site 1701), Saint Petersburg, Leningradskaya Oblast'
  - Federal Scientific Methodological AIDS Prevention and Control Center ( Site 1703), Moscow, Moscow
  - Infectious Clinical Hospital #2 ( Site 1719), Moscow, Moscow
  - FGU Republican Clinical Infectious Hospital of Roszdrav ( Site 1700), Saint Petersburg, Sankt-Peterburg
  - Regional Center for Prevent. and Control of AIDS and Inf. Diseases ( Site 1715), Yekaterinburg, Sverdlovsk Oblast
  - Republican Clinical Hospital of Infectious Diseases n. a. A.F.Agafonov ( Site 1707), Kazan', Tatarstan, Respublika
- South Africa (2):
  - JOSHA Research ( Site 1406), Bloemfontein, Free State
  - Desmond Tutu HIV Foundation Clinical Trial Unit ( Site 1414), Cape Town, Western Cape
- Spain (7):
  - Hospital General de Elche ( Site 1608), Elche, Alicante
  - Hospital Universitari Germans Trias i Pujol ( Site 1606), Badalona, Barcelona [Barcelona]
  - Hospital Clinic i Provincial ( Site 1600), Barcelona
  - Hospital General Universitario Gregorio Maranon ( Site 1603), Madrid
  - Hospital Universitario Infanta Leonor ( Site 1601), Madrid
  - Hospital Universitario Fundacion Jimenez Diaz ( Site 1602), Madrid
  - Hospital Universitario La Paz ( Site 1604), Madrid
- Switzerland (6):
  - Universitaetsspital Basel ( Site 3302), Basel, Canton of Basel-City
  - Inselspital Universitaetsspital Bern ( Site 3303), Bern, Canton of Bern
  - Hopitaux Universitaires de Geneve HUG. ( Site 3304), Geneva, Canton of Geneva
  - Kantonsspital St. Gallen ( Site 3301), Sankt Gallen, Canton of St. Gallen
  - Universitaetsspital Zuerich ( Site 3300), Zurich, Canton of Zurich
  - Ospedale Regionale di Lugano Civico ( Site 3305), Lugano, Canton Ticino
- United Kingdom (5):
  - Brighton and Sussex University Hospital NHS Trust ( Site 1908), Brighton, Brighton And Hove
  - Southmead Hospital ( Site 1910), Bristol, Bristol, City of
  - Royal Free Hospital ( Site 1904), London, Camden
  - Kings College Hospital NHS Foundation Trust ( Site 1907), London, London, City of
  - North Manchester General Hospital ( Site 1902), Manchester

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Molina JM, Rizzardini G, Orrell C, Afani A, Calmy A, Oka S, Hinestrosa F, Kumar P, Tebas P, Walmsley S, Grandhi A, Klopfer S, Gendrano I, Eves K, Correll TA, Fox MC, Kim J. Switch to fixed-dose doravirine (100 mg) with islatravir (0.75 mg) once daily in virologically suppressed adults with HIV-1 on antiretroviral therapy: 48-week results of a phase 3, randomised, open-label, non-inferiority trial. Lancet HIV. 2024 Jun;11(6):e369-e379. doi: 10.1016/S2352-3018(24)00031-6. Epub 2024 May 8. PMID 38734015
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Adult human immunodeficiency virus-1 (HIV-1)-infected participants receiving baseline antiretroviral therapy (ART) were enrolled. 672 participants were randomly assigned in a 1:1 ratio to either Group 1: participants switched from baseline ART to doravirine (DOR)/islatravir (ISL) on Day 1 to Week 96; or Group 2: participants continued baseline ART until Week 48 then delayed switch to DOR/ISL from Week 48 to Week 96.
Groups:
- Group 1: Doravirine/Islatravir (DOR/ISL): Participants who were previously treated with continuous baseline antiretroviral therapy (ART) received DOR/ISL, a fixed dose combination (FDC) of 100 mg doravirine (DOR)/0.75 mg islatravir (ISL) orally once daily for 96 weeks.
Period: Overall Study
Arm/Group | Group 1: Doravirine/Islatravir (DOR/ISL) | Group 2: Baseline Antiretroviral Therapy (ART)
Started | 336 | 336
Group 1 Participants Who Received DOR/ISL From 0-48 Weeks | 336 | 0
Group 1 Participants Who Received DOR/ISL From 48-96 Weeks | 322 | 0
Group 2 Participants Who Received Baseline ART From Weeks 0-48 | 0 | 336
Group 2 Participants Who Delayed Switch Over to DOR/ISL Weeks 48-96 | 0 | 326
Completed | 279 | 299
Not Completed | 57 | 37
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 4 | 5
Not completed — Physician Decision | 10 | 6
Not completed — Withdrawal by Subject | 35 | 17
Not completed — Not Reported | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Doravirine/Islatravir (DOR/ISL) | Group 2: Baseline Antiretroviral Therapy (ART) | Total
Number analyzed (Participants) | 336 | 336 | 672
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.5 (11.7) | 45.4 (11.7) | 45.5 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 126 | 249
  Male | 213 | 210 | 423
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 67 | 64 | 131
  Not Hispanic or Latino | 266 | 270 | 536
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 8 | 12
  Asian | 19 | 19 | 38
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 88 | 91 | 179
  White | 210 | 198 | 408
  More than one race | 13 | 16 | 29
  Unknown or Not Reported | 2 | 2 | 4
ART Regimen Stratification [Count of Participants; unit: Participants] — Participants were stratified into the following baseline ART regimen: (1) Protease inhibitor (PI)-containing regimens (including PI- and integrase strand transferase inhibitor [InSTI]-containing regimens); (2) InSTI-based regimens (non-PI containing regimens); (3) All other non-PI- and non-InSTI containing regimens.
  Participants
    PI-containing regimens (including PI- and InSTI-containing regimens) | 46 | 46 | 92
    InSTI-based regimens (non-PI containing regimens) | 174 | 174 | 348
    All other non-PI- and non-InSTI containing regimens | 116 | 116 | 232

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Human Immunodeficiency Virus (HIV)-1 Ribonucleic Acid (RNA) ≥50 Copies/mL at Week 48
Description: HIV-1 RNA levels in blood samples taken at each visit were measured by the Abbott RealTime polymerase chain reaction (PCR) assay with a reliable lower limit of quantification of 40 copies/mL. The percentage of participants with HIV-1 RNA ≥50 copies/mL at Week 48 is presented using the FDA Snapshot missing data approach.
Time Frame: Week 48
Population: All randomized participants who received at least one dose of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Doravirine/Islatravir (DOR/ISL) | Group 2: Baseline Antiretroviral Therapy (ART)
Number analyzed (Participants) | 336 | 336
Percentage of Participants | 0.0 | 1.5
Statistical Analysis 1: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Test type: Non-Inferiority — Doravirine/Islatravir (DOR/ISL) - Baseline Antiretroviral Therapy (ART). Non-inferiority was concluded if the upper bound of the 2-sided multiplicity-adjusted 95% CI was less than 4 percentage points; p < .001, Miettinen and Nurminen; The Miettinen and Nurminen method was stratified by corrected baseline ART regimen with Cochran-Mantel-Haenszel (CMH) weights; Estimated Difference = -1.49, 95% CI 2-sided [-3.44 to -0.34]

2. Primary Outcome: Percentage of Participants With One or More Adverse Events (AEs) up to Week 48
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experienced at least one AE was reported.
Time Frame: Up to ~48 Weeks
Population: All randomized participants who received at least one dose of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Doravirine/Islatravir (DOR/ISL) | Group 2: Baseline Antiretroviral Therapy (ART)
Number analyzed (Participants) | 336 | 336
Percentage of Participants | 80.1 | 70.2
Statistical Analysis 1: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Test type: Other — Difference in percentage versus Baseline Antiretroviral Therapy (ART). Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = 9.8, 95% CI 2-sided [3.3 to 16.3] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method

3. Primary Outcome: Percentage of Participants Who Discontinued Study Intervention Due to an AE up to Week 48
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who discontinued study intervention due to an AE was reported.
Time Frame: Up to ~48 Weeks
Population: All randomized participants who received at least one dose of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Doravirine/Islatravir (DOR/ISL) | Group 2: Baseline Antiretroviral Therapy (ART)
Number analyzed (Participants) | 336 | 336
Percentage of Participants | 2.1 | 0.3
Statistical Analysis 1: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Test type: Other — [test comment as in outcome 2, analysis 1]; Estimated Difference = 1.8, 95% CI 2-sided [0.2 to 4.0] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method

4. Secondary Outcome: Percentage of Participants With HIV-1 RNA <40 or <50 Copies/mL at Week 48
Description: HIV-1 RNA levels in blood samples taken at each visit were measured by the Abbott RealTime PCR assay with a reliable lower limit of quantification of 40 copies/mL. The percentage of participants with HIV-1 RNA <40 copies/mL or <50 copies/mL at Week 48 is presented using the FDA Snapshot missing data approach.
Time Frame: Week 48
Population: All randomized participants who received at least one dose of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Doravirine/Islatravir (DOR/ISL) | Group 2: Baseline Antiretroviral Therapy (ART)
Number analyzed (Participants) | 336 | 336
Percentage of Participants
  HIV-1 RNA <40 copies/mL | 94.6 | 94.3
  HIV-1 RNA <50 copies/mL | 95.2 | 94.3
Statistical Analysis 1: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); HIV-1 RNA <40 copies/mL; Test type: Other — Doravirine/Islatravir (DOR/ISL)- Baseline Antiretroviral Therapy (ART). Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = 0.30, 95% CI 2-sided [-3.28 to 3.90] — The Miettinen and Nurminen method was stratified by corrected baseline ART regimen with Cochran-Mantel-Haenszel (CMH) weights
Statistical Analysis 2: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); HIV-1 RNA <50 copies/mL; Test type: Other — [test comment as in outcome 4, analysis 1]; Estimated Difference = 0.89, 95% CI 2-sided [-2.58 to 4.43] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Group 2 (Switch-Over): Percentage of Participants With HIV-1 RNA ≥50 Copies/mL, <40 Copies/mL or <50 Copies/mL at Week 96
Description: HIV-1 RNA levels in blood samples taken at each visit was measured by the Abbott RealTime PCR assay with a reliable lower limit of quantification of 40 copies/mL. The percentage of participants with HIV-1 RNA ≥50 copies/mL, <40 copies/mL, or <50 copies/mL at Week 96 is reported for Group 2 participants who delayed switch over from baseline ART to DOR/ISL from Week 48 to Week 96. Per protocol, the percentage of participants with HIV-1 RNA ≥50 copies/mL, <40 copies/mL, or <50 copies/mL at Week 96 for Group 1 participants is a separate outcome measure and is presented later in the record.
Time Frame: Week 96
Population: The analysis population consisted of all randomized participants in Group 2 who delayed switch over from baseline ART to DOR/ISL from Week 48 to Week 96 who received at least one dose of study intervention and had data available for this outcome measure. Per protocol, the percentage of participants with HIV-1 RNA ≥50 copies/mL, <40 copies/mL, or <50 copies/mL at Week 96 for Group 1 participants is a separate outcome measure and is presented later in the record.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Group 1: Doravirine/Islatravir (DOR/ISL) | Group 2: Baseline Antiretroviral Therapy (ART)
Number analyzed (Participants) | 0 | 326
Percentage of Participants
  HIV-1 RNA ≥50 copies/mL |  | 0.9 [0.2 to 2.7]
  HIV-1 RNA <50 copies/mL |  | 89.6 [85.7 to 92.7]
  HIV-1 RNA <40 copies/mL |  | 89.6 [85.7 to 92.7]

6. Secondary Outcome: Group 1: Percentage of Participants With HIV-1 RNA ≥50 Copies/mL, <40 Copies/mL or <50 Copies/mL at Week 96
Description: HIV-1 RNA levels in blood samples taken at each visit was measured by the Abbott RealTime PCR assay with a reliable lower limit of quantification of 40 copies/mL. The percentage of participants with HIV-1 RNA ≥50 copies/mL, <40 copies/mL, or <50 copies/mL at Week 96 is reported for Group 1 participants. Per protocol, the percentage of participants with HIV-1 RNA ≥50 copies/mL, <40 copies/mL, or <50 copies/mL at Week 96 for Group 2 participants who delayed switch over from baseline ART to DOR/ISL from Week 48 to Week 96 is a separate outcome measure and is presented earlier in the record.
Time Frame: Week 96
Population: The analysis population consisted of all randomized participants in Group 1 who received at least one dose of study intervention and had data available for this outcome measure. Per protocol, the percentage of participants with HIV-1 RNA ≥50 copies/mL, <40 copies/mL, or <50 copies/mL at Week 96 for Group 2 participants who delayed switch over from baseline ART to DOR/ISL from Week 48 to Week 96 is a separate outcome measure and is presented earlier in the record.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Group 1: Doravirine/Islatravir (DOR/ISL) | Group 2: Baseline Antiretroviral Therapy (ART)
Number analyzed (Participants) | 336 | 0
Percentage of Participants
  HIV-1 RNA ≥50 copies/mL | 1.2 [0.3 to 3.0] |
  HIV-1 RNA <40 copies/mL | 86.0 [81.8 to 89.5] |
  HIV-1 RNA <50 copies/mL | 85.7 [81.5 to 89.3] |

7. Secondary Outcome: Percentage Change From Baseline in CD4+ T-cell Count at Week 48
Description: Plasma CD4+ T-Cell Count was measured in cells/mm^3 for baseline and 48 weeks. Baseline measurements were defined as the Day 1 value of each participant. The percentage change from baseline to Week 48 is presented.
Time Frame: Baseline and Week 48
Population: All randomized participants who received at least one dose of study intervention and who have baseline data.
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Group 1: Doravirine/Islatravir (DOR/ISL) | Group 2: Baseline Antiretroviral Therapy (ART)
Number analyzed (Participants) | 313 | 311
Percentage Change | -0.7 [-4.0 to 2.6] | 8.7 [5.4 to 12.0]
Statistical Analysis 1: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Test type: Other — [test comment as in outcome 2, analysis 1]; Estimated Difference = -8.9, 95% CI 2-sided [-13.4 to -4.5] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method

8. Secondary Outcome: Group 1: Percentage Change From Baseline in CD4+ T-cell Count at Week 96
Description: Plasma CD4+ T-Cell Count was measured in cells/mm^3 for baseline and 96 weeks. Baseline measurements were defined as the Day 1 value of each participant. The mean percent change from baseline to Week 96 in CD4+ T-cell count is reported for Group 1 participants. Per protocol, the mean percentage change from baseline in CD4+ T-cell count at Week 96 for Group 2 participants was not planned or conducted.
Time Frame: Baseline and Week 96
Population: The analysis population consisted of all randomized participants in Group 1 who received at least one dose of study intervention and had data, including baseline data, available for this outcome measure. Per protocol, the percentage change from baseline in CD4+ T-cell count at Week 96 for Group 2 participants was not planned or conducted.
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Group 1: Doravirine/Islatravir (DOR/ISL) | Group 2: Baseline Antiretroviral Therapy (ART)
Number analyzed (Participants) | 284 | 0
Percentage Change | 4.49 [0.56 to 8.43] |

9. Secondary Outcome: Group 1 & Group 2 (Switch-Over): Percentage Change From Week 48 in CD4+ T-cell Count at Week 96
Description: Plasma CD4+ T-Cell Count was measured in cells/mm^3 for Week 48 and Week 96. The mean percent change from Week 48 to Week 96 is reported for Group 1 and Group 2 participants who delayed switch over from baseline ART to DOR/ISL Week 48 to Week 96.
Time Frame: Week 48 and Week 96
Population: The analysis population consisted of all randomized participants who received at least one dose of study intervention and had data available for this outcome measure for participants in Group 1 and participants in Group 2 who delayed switch over from baseline ART to DOR/ISL from Week 48 to Week 96.
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Group 1: Doravirine/Islatravir (DOR/ISL) | Group 2: Baseline Antiretroviral Therapy (ART)
Number analyzed (Participants) | 289 | 285
Percentage Change | 5.29 [1.99 to 8.58] | 0.16 [-2.96 to 3.29]

10. Secondary Outcome: Percentage of Participants With Evidence of Viral Drug Resistance-associated Substitutions at Week 48
Description: Viral drug resistance is defined as participants with confirmed HIV-1 RNA ≥400 copies/mL and/or genotypic or phenotypic analysis of data showing evidence of resistance to the study drug administered. The percentage of participants who demonstrated drug resistance at Week 48 is presented.
Time Frame: Week 48
Population: Participants who met the definition of confirmed virologic rebound (two consecutive [2 to 4 weeks apart] occurrences of HIV-1 RNA ≥200 copies/mL) at any time during the study or who discontinued study intervention for another reason and have HIV-1 RNA ≥200 copies/mL at the time of discontinuation. Participants for whom available genotypic or phenotypic data showed evidence of resistance, irrespective of viral load, were also included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Doravirine/Islatravir (DOR/ISL) | Group 2: Baseline Antiretroviral Therapy (ART)
Number analyzed (Participants) | 336 | 336
Percentage of Participants | 0.0 | 0.9

11. Secondary Outcome: Percentage of Participants With Evidence of Viral Drug Resistance-associated Substitutions at Week 96
Description: Viral drug resistance was defined as participants with confirmed HIV-1 RNA ≥400 copies/mL and/or genotypic or phenotypic analysis of data showing evidence of resistance to the study drug administered. The percentage of participants who demonstrate drug resistance at Week 96 is presented for Group 1 and Group 2 participants who delayed switch over from baseline ART to DOR/ISL from Week 48 to Week 96. Per protocol, the percentage of participants with evidence of viral drug resistance-associated substitutions from week 0 to week 48 for Group 1 and Group 2 participants is a separate outcome measure and is presented earlier in the record.
Time Frame: Week 96
Population: Analysis population included participants with virologic rebound (2 repeated incidents of HIV-1 RNA ≥200 copies/mL, 2-4 weeks apart) or who discontinued study intervention with HIV-1 RNA ≥200 copies/mL. Participants with available data showing resistance, despite viral load, are included. Per protocol, percentage of participants with evidence of viral drug resistance associated substitutions from week 0 to week 48 for Groups 1 and 2 is a separate outcome measure reported earlier in the record.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Doravirine/Islatravir (DOR/ISL) | Group 2: Baseline Antiretroviral Therapy (ART)
Number analyzed (Participants) | 336 | 326
Percentage of Participants | 0.0 | 0.0

12. Secondary Outcome: Change From Baseline to Week 24 in Fasting Lipids in Participants on Protease Inhibitor (PI)-Containing Regimens (Including PI- and Integrase Strand Transferase Inhibitor [InSTI]-Containing Regimens)
Description: Blood serum samples were taken at baseline and Week 24. Per protocol, this outcome analysis was conducted in participants on PI-containing regimens (including PI- and InSTI-containing regimens), excluding participants who took lipid-lowering therapy during the study. The fasting lipids consisted of fasting cholesterol, fasting high density lipoprotein (HDL) cholesterol, fasting low density lipoprotein (LDL) cholesterol, fasting non-HDL cholesterol, and fasting triglycerides. The mean change from baseline to Week 24 in fasting lipids is presented.
Time Frame: Baseline and Week 24
Population: All randomized participants on PI-containing regimens (including PI- and InSTI-containing regimens) who received at least one dose of study intervention and had baseline and Week 24 data available for each lipid type, excluding participants who took lipid-lowering therapy during the study, per protocol.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Group 1: Doravirine/Islatravir (DOR/ISL) | Group 2: Baseline Antiretroviral Therapy (ART)
Number analyzed (Participants) | 32 | 40
mg/dL
  Fasting Cholesterol | -12.94 [-23.94 to -1.94] | 6.20 [-2.16 to 14.56]
  Fasting HDL | -0.97 [-5.94 to 4.00] | 0.76 [-1.80 to 3.32]
  Fasting LDL Cholesterol | -7.47 [-15.86 to 0.92] | 5.93 [-1.08 to 12.93]
  Fasting Non-HDL Cholesterol | -11.97 [-21.83 to -2.10] | 5.44 [-2.29 to 13.16]
  Fasting Triglycerides | -22.69 [-42.92 to -2.46] | -3.16 [-19.81 to 13.49]
Statistical Analysis 1: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting Cholesterol; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = -19.75, 95% CI 2-sided [-33.07 to -6.44] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method
Statistical Analysis 2: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting HDL Cholesterol; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = -1.35, 95% CI 2-sided [-6.55 to 3.84] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method
Statistical Analysis 3: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting LDL Cholesterol; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = -13.94, 95% CI 2-sided [-24.69 to -3.20] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method
Statistical Analysis 4: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting Non-HDL Cholesterol; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = -17.74, 95% CI 2-sided [-30.02 to -5.46] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method
Statistical Analysis 5: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting Triglycerides; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = -21.28, 95% CI 2-sided [-45.51 to 2.96] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method

13. Secondary Outcome: Change From Baseline to Week 24 in Fasting Lipids in Participants on InSTI-based Regimens (Non-PI Containing Regimens)
Description: Blood serum samples were taken at baseline and Week 24. Per protocol, this outcome analysis was conducted in participants on InSTI-based regimens (non-PI containing regimens), excluding participants who took lipid-lowering therapy during the study. The fasting lipids consisted of fasting cholesterol, fasting HDL cholesterol, fasting LDL cholesterol, fasting non-HDL cholesterol, and fasting triglycerides. The mean change from baseline to Week 24 in fasting lipids is presented.
Time Frame: Baseline and Week 24
Population: All randomized participants on InSTI-based regimens (non-PI containing regimens) who received at least one dose of study intervention and had baseline and Week 24 data available for each lipid type, excluding participants who took lipid-lowering therapy during the study, per protocol.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Group 1: Doravirine/Islatravir (DOR/ISL) | Group 2: Baseline Antiretroviral Therapy (ART)
Number analyzed (Participants) | 130 | 135
mg/dL
  Fasting Cholesterol | 2.98 [-2.19 to 8.14] | 8.74 [4.25 to 13.23]
  Fasting HDL Cholesterol | 0.84 [-1.11 to 2.79] | 0.27 [-1.06 to 1.60]
  Fasting LDL Cholesterol: number analyzed (Participants) | 128 | 135
  Fasting LDL Cholesterol | 3.21 [-1.49 to 7.92] | 8.50 [4.27 to 12.73]
  Fasting Non-HDL Cholesterol | 2.14 [-3.39 to 7.67] | 8.47 [4.05 to 12.90]
  Fasting Triglycerides | -0.97 [-17.98 to 16.04] | -1.56 [-10.80 to 7.69]
Statistical Analysis 1: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting Cholesterol; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = -4.17, 95% CI 2-sided [-10.43 to 2.09] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method
Statistical Analysis 2: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting HDL Cholesterol; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = 0.81, 95% CI 2-sided [-1.46 to 3.09] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method
Statistical Analysis 3: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting LDL Cholesterol; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = -3.87, 95% CI 2-sided [-9.47 to 1.74] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method
Statistical Analysis 4: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting Non-HDL Cholesterol; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = -4.92, 95% CI 2-sided [-11.21 to 1.38] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method
Statistical Analysis 5: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting Triglycerides; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = 1.65, 95% CI 2-sided [-16.14 to 19.43] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method

14. Secondary Outcome: Change From Baseline to Week 24 in Fasting Lipids in Participants on All Other Non-PI- and Non-InSTI Containing Regimens
Description: Blood serum samples were taken at baseline and Week 24. Per protocol, this outcome analysis was conducted in participants on all other non-PI- and non-InSTI containing regimens, excluding participants who took lipid-lowering therapy during the study. The fasting lipids consisted of fasting cholesterol, fasting HDL cholesterol, fasting LDL cholesterol, fasting non-HDL cholesterol, and fasting triglycerides. The mean change from baseline to Week 24 in fasting lipids is presented.
Time Frame: Baseline and Week 24
Population: All randomized participants on all other non-PI- and non-InSTI containing regimens, who received at least one dose of study intervention and had baseline and Week 24 data available for each lipid type, excluding participants who took lipid-lowering therapy during the study, per protocol.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Group 1: Doravirine/Islatravir (DOR/ISL) | Group 2: Baseline Antiretroviral Therapy (ART)
Number analyzed (Participants) | 89 | 95
mg/dL
  Fasting Cholesterol | 7.18 [-0.49 to 14.85] | 7.35 [2.44 to 12.25]
  Fasting HDL Cholesterol: number analyzed (Participants) | 88 | 95
  Fasting HDL Cholesterol | -3.43 [-6.51 to -0.36] | -0.72 [-3.02 to 1.58]
  Fasting LDL Cholesterol: number analyzed (Participants) | 87 | 95
  Fasting LDL Cholesterol | 11.33 [5.75 to 16.92] | 7.19 [3.35 to 11.04]
  Fasting Non-HDL Cholesterol: number analyzed (Participants) | 88 | 95
  Fasting Non-HDL Cholesterol | 11.07 [4.40 to 17.74] | 8.07 [4.10 to 12.04]
  Fasting Triglycerides: number analyzed (Participants) | 88 | 95
  Fasting Triglycerides | -1.16 [-14.27 to 11.95] | 4.45 [-3.89 to 12.80]
Statistical Analysis 1: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting Cholesterol; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = 1.05, 95% CI 2-sided [-7.60 to 9.70] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method
Statistical Analysis 2: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting HDL Cholesterol; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = -3.16, 95% CI 2-sided [-6.37 to 0.05] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method
Statistical Analysis 3: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting LDL Cholesterol; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = 4.38, 95% CI 2-sided [-2.27 to 11.03] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method
Statistical Analysis 4: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting Non-HDL Cholesterol; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = 3.63, 95% CI 2-sided [-3.93 to 11.19] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method
Statistical Analysis 5: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting Triglycerides; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = -1.79, 95% CI 2-sided [-15.89 to 12.31] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method

15. Secondary Outcome: Change From Baseline to Week 48 in Fasting Lipids in Participants on Protease Inhibitor (PI)-Containing Regimens (Including PI- and Integrase Strand Transferase Inhibitor [InSTI]-Containing Regimens)
Description: Blood serum samples were taken at baseline and Week 48. Per protocol, this outcome analysis was conducted in participants on PI-containing regimens (including PI- and InSTI-containing regimens), excluding participants who took lipid-lowering therapy during the study. The fasting lipids consisted of fasting cholesterol, fasting high density lipoprotein (HDL) cholesterol, fasting low density lipoprotein (LDL) cholesterol, fasting non-HDL cholesterol, and fasting triglycerides. The mean change from baseline to Week 48 in fasting lipids is presented.
Time Frame: Baseline and Week 48
Population: All randomized participants on PI-containing regimens (including PI- and InSTI-containing regimens) who received at least one dose of study intervention and had baseline and Week 48 data available for each lipid type, excluding participants who took lipid-lowering therapy during the study, per protocol.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Group 1: Doravirine/Islatravir (DOR/ISL) | Group 2: Baseline Antiretroviral Therapy (ART)
Number analyzed (Participants) | 29 | 37
mg/dL
  Fasting Cholesterol | -15.31 [-28.99 to -1.64] | 1.84 [-5.70 to 9.38]
  Fasting HDL Cholesterol: number analyzed (Participants) | 29 | 36
  Fasting HDL Cholesterol | -1.45 [-6.01 to 3.11] | -1.08 [-3.91 to 1.75]
  Fasting LDL Cholesterol: number analyzed (Participants) | 29 | 35
  Fasting LDL Cholesterol | -8.59 [-19.72 to 2.54] | 3.37 [-3.30 to 10.04]
  Fasting Non-HDL Cholesterol: number analyzed (Participants) | 29 | 36
  Fasting Non-HDL Cholesterol | -13.86 [-25.28 to -2.45] | 2.81 [-4.40 to 10.01]
  Fasting Triglycerides: number analyzed (Participants) | 29 | 36
  Fasting Triglycerides | -26.90 [-42.31 to -11.48] | 2.28 [-16.39 to 20.95]
Statistical Analysis 1: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting Cholesterol; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = -18.41, 95% CI 2-sided [-32.05 to -4.76] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method
Statistical Analysis 2: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting HDL Cholesterol; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = 0.01, 95% CI 2-sided [-5.06 to 5.08] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method
Statistical Analysis 3: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting LDL Cholesterol; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = -14.12, 95% CI 2-sided [-25.81 to -2.43] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method
Statistical Analysis 4: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting Non-HDL Cholesterol; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = -18.23, 95% CI 2-sided [-30.45 to -6.00] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method
Statistical Analysis 5: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting Triglycerides; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = -27.79, 95% CI 2-sided [-51.08 to -4.49] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method
Statistical Analysis 6: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting LDL Cholesterol - Multiplicity Adjusted; Test type: Superiority — Treatment Difference vs Baseline ART. Superiority will be concluded if the upper bound of the 2-sided multiplicity-adjusted 95% CI is less than 0 percentage points; p = 0.0094, ANCOVA — The significance level in ANCOVA model was 0.02497/2=0.012485. The p-value is statistically significant if it is <0.02497/2=0.012485; Mean Difference (Net) = -14.12, 95% CI 2-sided [-27.56 to -0.68]; The multiplicity adjusted 95% CIs for treatment difference were calculated from ANCOVA models with terms for baseline measurement and treatment
Statistical Analysis 7: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting Non-HDL Cholesterol - Multiplicity Adjusted; Test type: Superiority — [test comment as in outcome 15, analysis 6]; p = 0.0021, ANCOVA — [p-value comment as in outcome 15, analysis 6]; Mean Difference (Net) = -18.23, 95% CI 2-sided [-32.28 to -4.17]; [other analysis details as in outcome 15, analysis 6]

16. Secondary Outcome: Change From Baseline to Week 48 in Fasting Lipids in Participants on InSTI-based Regimens (Non-PI Containing Regimens)
Description: Blood serum samples were taken at baseline and Week 48. Per protocol, this outcome analysis was conducted in participants on InSTI-based regimens (non-PI containing regimens), excluding participants who took lipid-lowering therapy during the study. The fasting lipids consisted of fasting cholesterol, fasting HDL cholesterol, fasting LDL cholesterol, fasting non-HDL cholesterol, and fasting triglycerides. The mean change from baseline to Week 48 in fasting lipids is presented.
Time Frame: Baseline and Week 48
Population: All randomized participants on InSTI-based regimens (non-PI containing regimens) who received at least one dose of study intervention and had baseline and Week 48 data available for each lipid type, excluding participants who took lipid-lowering therapy during the study, per protocol.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Group 1: Doravirine/Islatravir (DOR/ISL) | Group 2: Baseline Antiretroviral Therapy (ART)
Number analyzed (Participants) | 129 | 137
mg/dL
  Fasting Cholesterol | 2.23 [-2.70 to 7.17] | 4.39 [-0.19 to 8.96]
  Fasting HDL Cholesterol: number analyzed (Participants) | 129 | 136
  Fasting HDL Cholesterol | 0.23 [-1.61 to 2.08] | 0.13 [-1.24 to 1.51]
  Fasting LDL Cholesterol: number analyzed (Participants) | 129 | 133
  Fasting LDL Cholesterol | 2.74 [-1.27 to 6.76] | 3.44 [-0.88 to 7.76]
  Fasting Non-HDL Cholesterol: number analyzed (Participants) | 129 | 136
  Fasting Non-HDL Cholesterol | 2.00 [-3.16 to 7.16] | 4.37 [-0.24 to 8.98]
  Fasting Triglycerides: number analyzed (Participants) | 129 | 136
  Fasting Triglycerides | -2.29 [-15.02 to 10.44] | 4.44 [-5.60 to 14.48]
Statistical Analysis 1: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting Cholesterol; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = -0.04, 95% CI 2-sided [-6.26 to 6.18] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method
Statistical Analysis 2: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting HDL Cholesterol; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = 0.35, 95% CI 2-sided [-1.84 to 2.54] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method
Statistical Analysis 3: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting LDL Cholesterol; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = 0.64, 95% CI 2-sided [-4.83 to 6.11] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method
Statistical Analysis 4: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting Non-HDL Cholesterol; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = -0.49, 95% CI 2-sided [-6.81 to 5.83] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method
Statistical Analysis 5: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting Triglycerides; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = -5.45, 95% CI 2-sided [-20.46 to 9.57] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method
Statistical Analysis 6: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting LDL Cholesterol - Multiplicity Adjusted; Test type: Superiority — [test comment as in outcome 15, analysis 6]; p = 0.4093, ANCOVA — [p-value comment as in outcome 15, analysis 6]; Mean Difference (Net) = 0.64, 95% CI 2-sided [-5.63 to 6.90]; [other analysis details as in outcome 15, analysis 6]
Statistical Analysis 7: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting Non-HDL Cholesterol - Multiplicity Adjusted; Test type: Superiority — [test comment as in outcome 15, analysis 6]; p = 0.4397, ANCOVA — [p-value comment as in outcome 15, analysis 6]; Mean Difference (Net) = -0.49, 95% CI 2-sided [-7.72 to 6.75]; [other analysis details as in outcome 15, analysis 6]

17. Secondary Outcome: Change From Baseline to Week 48 in Fasting Lipids in Participants on All Other Non-PI- and Non-InSTI Containing Regimens
Description: Blood serum samples were taken at baseline and Week 48. Per protocol, this outcome analysis was conducted in participants on all other non-PI- and non-InSTI containing regimens, excluding participants who took lipid-lowering therapy during the study. The fasting lipids consisted of fasting cholesterol, fasting HDL cholesterol, fasting LDL cholesterol, fasting non-HDL cholesterol, and fasting triglycerides. The mean change from baseline to Week 48 in fasting lipids is presented.
Time Frame: Baseline and Week 48
Population: All randomized participants on all other non-PI- and non-InSTI containing regimens, who received at least one dose of study intervention and had baseline and Week 48 data available for each lipid type, excluding participants who took lipid-lowering therapy during the study, per protocol.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Group 1: Doravirine/Islatravir (DOR/ISL) | Group 2: Baseline Antiretroviral Therapy (ART)
Number analyzed (Participants) | 91 | 95
mg/dL
  Fasting Cholesterol | 5.66 [-1.38 to 12.70] | 4.62 [0.10 to 9.15]
  Fasting HDL Cholesterol: number analyzed (Participants) | 90 | 95
  Fasting HDL Cholesterol | -3.84 [-6.72 to -0.97] | -1.98 [-4.60 to 0.63]
  Fasting LDL Cholesterol: number analyzed (Participants) | 90 | 94
  Fasting LDL Cholesterol | 9.27 [4.05 to 14.49] | 7.30 [3.97 to 10.63]
  Fasting Non-HDL Cholesterol: number analyzed (Participants) | 90 | 95
  Fasting Non-HDL Cholesterol | 9.94 [4.16 to 15.73] | 6.61 [3.13 to 10.08]
  Fasting Triglycerides: number analyzed (Participants) | 90 | 95
  Fasting Triglycerides | 3.33 [-9.54 to 16.21] | -2.97 [-12.37 to 6.43]
Statistical Analysis 1: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting Cholesterol; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = 2.31, 95% CI 2-sided [-5.54 to 10.17] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method
Statistical Analysis 2: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting HDL Cholesterol; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = -2.52, 95% CI 2-sided [-5.69 to 0.65] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method
Statistical Analysis 3: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting LDL Cholesterol; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = 2.34, 95% CI 2-sided [-3.73 to 8.42] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method
Statistical Analysis 4: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting Non-HDL Cholesterol; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = 3.97, 95% CI 2-sided [-2.63 to 10.56] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method
Statistical Analysis 5: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Fasting Triglycerides; Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = 10.50, 95% CI 2-sided [-3.97 to 24.96] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method

18. Secondary Outcome: Change From Baseline in Body Weight at Week 48 for InSTI-based Regimens (Non-PI-containing Regimens)
Description: Baseline measurements were defined as the Day 1 value of each participant. The change from baseline in body weight to Week 48 is presented for participants who received InSTI- based regimens.
Time Frame: Baseline and Week 48
Population: All randomized participants who received at least one dose of study intervention, had baseline and Week 48 data available for body weight, and received InSTI-based regimens.
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Group 1: Doravirine/Islatravir (DOR/ISL) | Group 2: Baseline Antiretroviral Therapy (ART)
Number analyzed (Participants) | 167 | 169
kg | 0.66 [-0.17 to 1.48] | 0.10 [-0.56 to 0.75]
Statistical Analysis 1: Comparison: Group 1: Doravirine/Islatravir (DOR/ISL) vs Group 2: Baseline Antiretroviral Therapy (ART); Test type: Other — Treatment Difference vs Baseline ART. Type of statistical test 'other' denotes no hypothesis testing was conducted; Estimated Difference = 0.44, 95% CI 2-sided [-0.59 to 1.46] — Difference in percentage versus (vs) Baseline ART was based on Miettinen & Nurminen method

19. Secondary Outcome: Group 1: Percentage of Participants With One or More AEs up to Week 96
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experienced at least one AE up to Week 96 is reported for Group 1 participants. Per protocol, the percentage of participants with one or more AEs for Group 2 participants is a separate outcome measure and is presented later in the record.
Time Frame: Up to ~96 Weeks
Population: The analysis population consisted of all randomized participants in Group 1 who received at least one dose of study intervention. Per protocol, the percentage of participants with one or more AEs for Group 2 participants is a separate outcome measure and is presented later in the record.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Doravirine/Islatravir (DOR/ISL) | Group 2: Baseline Antiretroviral Therapy (ART)
Number analyzed (Participants) | 336 | 0
Percentage of Participants | 92.3 |

20. Secondary Outcome: Group 1: Percentage of Participants Who Discontinued Study Intervention Due to an AE up to Week 96
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who discontinued study intervention due to an AE up to Week 96 is reported for Group 1 participants. Per protocol, the percentage of participants who discontinued study intervention for Group 2 participants is a separate outcome measure and is presented later in the record.
Time Frame: Up to ~96 Weeks
Population: The analysis population consisted of all randomized participants in Group 1 who received at least one dose of study intervention. Per protocol, the percentage of participants who discontinued study intervention for Group 2 participants is a separate outcome measure and is presented later in the record.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Doravirine/Islatravir (DOR/ISL) | Group 2: Baseline Antiretroviral Therapy (ART)
Number analyzed (Participants) | 336 | 0
Percentage of Participants | 5.7 |

21. Secondary Outcome: Group 1 & Group 2 (Switch-Over): Percentage of Participants With One or More AEs From Week 48 to Week 96
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experienced at least one AE from Week 48 up to Week 96 is reported for Group 1 participants and Group 2 participants who delayed switch over from baseline ART to DOR/ISL from Week 48 to Week 96.
Time Frame: Weeks 48-96 (up to ~48 weeks)
Population: The analysis population consisted of all randomized participants who received at least one dose of study intervention for participants in Group 1 and participants in Group 2 who delayed switch over from baseline ART to DOR/ISL from Week 48 to Week 96.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Doravirine/Islatravir (DOR/ISL) | Group 2: Baseline Antiretroviral Therapy (ART)
Number analyzed (Participants) | 322 | 326
Percentage of Participants | 73.0 | 76.4

22. Secondary Outcome: Group 1 & Group 2 (Switch-Over): Percentage of Participants Who Discontinued Study Intervention Due to an AE From Week 48 to Week 96
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who discontinued study intervention due to an AE from Week 48 up to Week 96 is reported for Group 1 participants and Group 2 participants who delayed switch over from baseline ART to DOR/ISL from Week 48 to Week 96.
Time Frame: Weeks 48-96 (up to ~48 weeks)
Population: as for outcome 21
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Doravirine/Islatravir (DOR/ISL) | Group 2: Baseline Antiretroviral Therapy (ART)
Number analyzed (Participants) | 322 | 326
Percentage of Participants | 3.7 | 2.5

ADVERSE EVENTS:
Time Frame: Up to approximately 49 months
Description: All-cause mortality (ACM): all randomized participants; AEs: all randomized participants who received at least one dose of study treatment. ACM and AEs have been reported separately for Weeks 0-48 and Weeks 48 - End of Trial. Per protocol, pregnancy-related AEs, and infant serious adverse events were collected on pregnant participants enrolled in the study. They are included by the arms in which the participants were enrolled.
Groups:
- Group 1: DOR/ISL Weeks 0-48; Group 1: DOR/ISL Weeks 48-End of Trial: Participants who were previously treated with continuous baseline antiretroviral therapy (ART) received DOR/ISL, a fixed dose combination (FDC) of 100 mg doravirine (DOR)/0.75 mg islatravir (ISL) orally once daily for 96 weeks.
- Group 2: Baseline ART Weeks 0-48; Group 2: DOR/ISL Weeks 48-End of Trial: Participants received continuous baseline ART for 48 weeks. Continuing participants delayed switch over from baseline ART to DOR/ISL, fixed dose combination of 100 mg DOR/0.75 mg ISL orally once daily, from Week 48 to Week 96, a total DOR/ISL treatment duration of 48 Weeks.
Arm/Group | Group 1: DOR/ISL Weeks 0-48 | Group 1: DOR/ISL Weeks 48-End of Trial | Group 2: Baseline ART Weeks 0-48 | Group 2: DOR/ISL Weeks 48-End of Trial
All-Cause Mortality (participants affected / at risk) | 0/336 | 1/322 | 1/336 | 0/326
Serious Adverse Events (participants affected / at risk) | 16/336 | 13/322 | 15/336 | 12/326
Other Adverse Events (participants affected / at risk) | 85/336 | 115/322 | 52/336 | 120/326
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: DOR/ISL Weeks 0-48 (N=336) | Group 1: DOR/ISL Weeks 48-End of Trial (N=322) | Group 2: Baseline ART Weeks 0-48 (N=336) | Group 2: DOR/ISL Weeks 48-End of Trial (N=326)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Omphalitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritoneal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Plasmodium falciparum infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy neonatal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuralgic amyotrophy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paranoia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: DOR/ISL Weeks 0-48 (N=336) | Group 1: DOR/ISL Weeks 48-End of Trial (N=322) | Group 2: Baseline ART Weeks 0-48 (N=336) | Group 2: DOR/ISL Weeks 48-End of Trial (N=326)
COVID-19 (Infections and infestations) | 18 (19) | 42 (42) | 15 (16) | 57 (60)
Accidental overdose (Injury, poisoning and procedural complications) | 24 (28) | 4 (4) | 3 (4) | 8 (12)
CD4 lymphocytes decreased (Investigations) | 2 (2) | 45 (47) | 0 (0) | 39 (41)
Lymphocyte count decreased (Investigations) | 0 (0) | 65 (70) | 0 (0) | 44 (46)
Osteopenia (Musculoskeletal and connective tissue disorders) | 10 (10) | 2 (2) | 19 (19) | 7 (7)
Headache (Nervous system disorders) | 36 (41) | 12 (14) | 16 (17) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/78/NCT04223778/Prot_SAP_001.pdf